CLINICAL TRIAL: NCT02363166
Title: Molecular Epidemiology and Phylodynamic and Phylogeographic Analysis of Community-associated Methicillin-resistant Staphylococcus Aureus (CA-MRSA) Transmission: An Emergency Department Population Sampling Strategy
Brief Title: Analysis of CA-MRSA Transmission: An ED Population Sampling Strategy
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: IRB201400426
Record Dates: First submitted 2015-02-09; First posted 2015-02-13 (Estimated); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Methicillin-Resistant Staphylococcus Aureus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Genomic DNA (gDNA) will be isolated from pelleted bacteria using the Roche High Pure PCR kit following the standard protocol for isolation of nucleic acids from bacteria. The quality of the extracted gDNA will be determined through gel electrophoresis and the quantity through Nanodrop2000.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Acute Abscess Group: Adults and pediatric patients presenting to the UFHealth Shands Emergency Department with evidence of an acute abscess, or skin/soft tissue infection, which can be sampled for culture and sensitivity testing will be recruited.
  Interventions: Other: Acute Abscess Group

INTERVENTIONS:
Other: Acute Abscess Group — Samples collected for culture and sensitivity testing depending on acute abscess, or skin/soft tissue infection.

SUMMARY:
Given that the Emergency Department (ED) has become the entry way for large populations of patients into the health care system, a strategy of sampling MRSA isolates in ED populations and merging this information with patient-level data may present a window to hypothesize and investigate CA-MRSA transmission within the community and its impact on hospital-acquired infections.

DETAILED DESCRIPTION:
Prospective cross-sectional study involving 500 patients enrolled over a one year period at the UFHealth Shands Hospital's Adult and Pediatric Emergency Department. The collected information will serve as pilot data for a future large comprehensive multi-site study.

Patients will have a wound culture and a nasal swab obtained as part of the study, which will be assessed for MRSA isolates using next-generation whole genome sequencing. The principal investigator or PI designee will also survey participants and review hospital records.

ELIGIBILITY:
Inclusion Criteria:

* Patient or Legally Authorized Representative (LAR) must have voluntarily signed an Institutional Review Board-approved informed consent form before initiation of any study procedures
* Patient presents with an acute abscess or a non-post-operative skin/soft tissue infection
* Patient presents through the UFHealth Shands Emergency Department

Exclusion Criteria:

* Patients who are employed by UFHealth and provide direct patient care
* Patients who have previously been enrolled in the study
* Patients who are not suitable for the study in the opinion of the investigator

Min Age: 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adult and pediatric patients presenting to the UFHealth Shands Emergency Department with evidence of an acute abscess, or skin/soft tissue infection (SSTI), which can be sampled for culture and sensitivity testing
Sampling Method: Non-Probability Sample
Enrollment: 575 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2018-04-04 (Actual); Study Completion 2018-04-04 (Actual)

PRIMARY OUTCOMES:
Strain Relatedness Identification Through Phylogenetic Analysis | 1 Hour
  Molecular (spa-typing) and genomic (WGS) relatedness of MRSA strains in isolates in ED populations presenting with SSTIs.

SECONDARY OUTCOMES:
Strain Transmission Through Analysis of Genetic Clustering | 1 year
  Phlyodynamic analysis of MRSA transmission course by strain
Patient Level Characteristics of Skin and Soft Tissue Infection (SSTI) Presentation | 6 Months
  To determine patient-level characteristics, including social and medical history, associated with a presentation related to SSTIs.
Pediatric and Adult Population Presentation Characteristics in Skin and Soft Tissue Infection (SSTI) | 6 Months
  Compare patient-level characteristics and phylogenetic clustering between pediatric and adult patients presenting with SSTIs.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph A Tyndall, MD, Principal Investigator — University of Florida
Locations (1):
- UF Health, Gainesville, Florida, United States

REFERENCES:
- [Background] Burton DC, Edwards JR, Horan TC, Jernigan JA, Fridkin SK. Methicillin-resistant Staphylococcus aureus central line-associated bloodstream infections in US intensive care units, 1997-2007. JAMA. 2009 Feb 18;301(7):727-36. doi: 10.1001/jama.2009.153. PMID 19224749
- [Background] Climo MW. Decreasing MRSA infections: an end met by unclear means. JAMA. 2009 Feb 18;301(7):772-3. doi: 10.1001/jama.2009.149. No abstract available. PMID 19224756
- [Background] Prosperi M, Veras N, Azarian T, Rathore M, Nolan D, Rand K, Cook RL, Johnson J, Morris JG Jr, Salemi M. Molecular epidemiology of community-associated methicillin-resistant Staphylococcus aureus in the genomic era: a cross-sectional study. Sci Rep. 2013;3:1902. doi: 10.1038/srep01902. PMID 23712667
- [Background] Park SH, Park C, Yoo JH, Choi SM, Choi JH, Shin HH, Lee DG, Lee S, Kim J, Choi SE, Kwon YM, Shin WS. Emergence of community-associated methicillin-resistant Staphylococcus aureus strains as a cause of healthcare-associated bloodstream infections in Korea. Infect Control Hosp Epidemiol. 2009 Feb;30(2):146-55. doi: 10.1086/593953. PMID 19128184
- [Background] Wu D, Wang Q, Yang Y, Geng W, Wang Q, Yu S, Yao K, Yuan L, Shen X. Epidemiology and molecular characteristics of community-associated methicillin-resistant and methicillin-susceptible Staphylococcus aureus from skin/soft tissue infections in a children's hospital in Beijing, China. Diagn Microbiol Infect Dis. 2010 May;67(1):1-8. doi: 10.1016/j.diagmicrobio.2009.12.006. Epub 2010 Mar 12. PMID 20227225